CLINICAL TRIAL: NCT02433899
Title: A Clinical Comparison of Microsurgical Versus Conventional Surgical Approaches for the Semilunar Coronally Advanced Flap
Brief Title: Microsurgical Versus Conventional Semilunar Coronally Advanced Flap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP CMM/HUAP no 162/2010
Record Dates: First submitted 2015-01-08; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Microsurgery; Dexamethasone; chlorhexidine gluconate; Mepivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test - Microsurgical semilunar flap (Experimental): Semilunar coronally repositioned flap performed under magnification with a surgical microscope.
  SLI was carried out following the outline of the gingival margin with a microsurgical blade under (8x) magnification. An ISI was performed mid-facially. Then, a split-thickness dissection was performed from the initial incision coronally until connecting to the ISI. The mid-facial tissue was completely released, positioned coronally to the CEJ and held in place against the tooth. A cyanoacrilate adhesive (CAA) was applied over the post-surgical gingival margin and tooth enamel to stabilize the flap.
  Interventions: Procedure: MICROSURGERY; Drug: Dexamethasone; Drug: Chlorhexidine gluconate; Drug: 2.0% Mepivacaine + 1:100.000 epinephrine
- Control - Conventional Semilunar flap (Active Comparator): Semilunar coronally repositioned flap performed without magnification. A semilunar incision (SLI) was carried out with a 15c surgical blade. An ISI was performed mid-facially. Then, a split-thickness dissection was performed from the initial incision coronally until connecting to the ISI. The mid-facial tissue was completely released, positioned coronally to the CEJ and held in place against the tooth. A cyanoacrilate adhesive (CAA) was applied over the post-surgical gingival margin and tooth enamel to stabilize the flap.
  Interventions: Procedure: MACROSURGERY; Drug: Dexamethasone; Drug: Chlorhexidine gluconate; Drug: 2.0% Mepivacaine + 1:100.000 epinephrine

INTERVENTIONS:
Procedure: MICROSURGERY — Semilunar coronally repositioned flap performed under magnification with a surgical microscope
  Other Names: Microsurgical semilunar flap
  Arms: Test - Microsurgical semilunar flap
Procedure: MACROSURGERY — Semilunar coronally repositioned flap performed without magnification
  Other Names: Original semilunar flap
  Arms: Control - Conventional Semilunar flap
Drug: Dexamethasone — 8mg Dexamethasone, single dose, 1 hour before surgery
Drug: Chlorhexidine gluconate — Oral rinses with chlorhexidine gluconate, BID, for 14 days
  Other Names: Gengilacer, LACER
Drug: 2.0% Mepivacaine + 1:100.000 epinephrine — Regional block
  Other Names: Mepiadre

SUMMARY:
BACKGROUND: The semilunar coronally repositioned flap (SLCRF) has been used for the treatment of recession defects (GR). Recently a microsusgical (MICRO) has been successfully employed with the procedure apparently resulting in improved results, however, no previous controlled clinical study has evaluated the MICRO SLCRF in comparison with SLCRF performed as originally described (MACRO). The objective of the present study was to compare the clinical outcomes of the MICRO and MACRO SLCRF in the treatment of human GR.

METHODS: Fourteen patients, with bilateral Miller class I GR defects were randomly assigned to MICRO or MACRO SLCRF. Clinical parameters, assessed at baseline and 6 months later, included recession height (RECH), recession width (RECW), width of keratinized tissue (WKT), probing depth (PD), clinical attachment level (CAL), pain measurements and esthetic evaluation with the Root Coverage Score (RCS). Inter-measurements differences were analyzed with a Chi-square or a paired t-test, with significance set at α<0.05.

DETAILED DESCRIPTION:
Study Population and Experimental Design The study was designed as a randomized, prospective, split-mouth, controlled clinical trial. It was conducted in accordance with the guidelines of the Helsinki Declaration of 1975, as revised in 2000, and after approved by institutional review board approval (CEP CMM/HUAP no 162/2010). Written informed consent was obtained from all patients after thorough explanation of the nature, risks, and benefits of the clinical investigation and associated procedures.

The study population consisted of patients referred for periodontal treatment at the School of Dentistry, Veiga de Almeida University, Brazil. In order to be elegible for the present study, adult individuals met the following inclusion criteria:

1. presence of bilateral Miller class I gingival recessions (≤ 3mm)
2. at least 2mm of keratinized tissue width (WKT)
3. endodontically-vital
4. maxillary canines or premolars.
5. shallow (<3mm) probing depth (PD)
6. no bleeding on probing.
7. absence of contraindications for periodontal surgery
8. no medications known to interfere with periodontal tissue health or healing
9. teeth to be treated free of caries or restorations

Exclusion criteria were:

1. presence of untreated periodontal disease
2. smokers
3. subjects with immunosuppressive systemic diseases (i.e., cancer, AIDS, diabetes)
4. Miller class II, III or class IV recession defects,
5. presence of apical radiolucency or caries or restorations in the areas to be treated,
6. previous lack of cooperation with the maintenance program

Fourteen patients (8 females and 6 males), 25 to 41 years of age (mean age, 31.6 years), were included in the study from January 2010 to December 2010. The primary outcome variable of the study was the reduction of recession depth. Sample size was determined by Power analysis, assuming α of .05, and a standard deviation of 0.7. This calculation indicated that with a sample of 14 subjects, the study would have >95% power to detect a 1-mm difference in recession depth between the two groups.

All patients were subjected to initial periodontal therapy 28 days before the beginning of the study. Treatment included oral hygiene instructions, scaling and root planning where needed, tooth polishing, plaque control measures and correction of traumatic tooth brushing technique. All patients were instructed and trained to use a soft toothbrush and to eliminate habits related to the etiology of the recession. Baseline full mouth plaque and bleeding scores were low. Each defect was randomly assigned to one of the two treatment modalities employed: (a) Controls (n=14): semilunar coronally repositioned flap performed without the aid of visual magnification (MACRO); (b) Test (n=14): SLCRF performed under magnification with a surgical microscope (MACRO) by the toss of a coin immediately before the surgical procedures, which were performed at the same clinical appointment. Single recession defects in 6 canines, 14 first-premolars, and 8 second-premolars were treated. Patients were not informed the site allocation for the surgical procedures.

Clinical data collection Clinical parameters were assessed and all measurements were recorded by a blinded, trained and calibrated examiner (ATD), unaware of the treatment provided, at baseline and 6 months later. Visual plaque score (VPS) and bleeding on probing (BOP) were assessed dichotomously at the mid-buccal location. Recession height (RECH) was measured as the distance from the CEJ to GM. Recession width (RECW) was measured as distance between the lateral borders of the recession at the level of the CEJ. The width of keratinized tissue (WKT) was measured as the distance between the GM and the MGJ. Thickness of the gingival tissues (GT) was measured 2mm apically to GM. PD was measured as the distance from the GM to the bottom of the gingival sulcus. PD and RECH were used to calculate the clinical attachment level (CAL). Measurements for PD and CAL were performed using an UNC #15 periodontal probe. Measurements of RECH, RECW, WKT and GT were performed with an endodontic spreader and rubber stopper (Maillefer, Dentsply, Brasil), and data was acquired with a digital gauge with 0.01mm resolution (Mitutoyo South America, Susano, Brazil).

Aesthetic and patient-related evaluations

Esthetic outcomes were evaluated with the Root Coverage Score (RCS) (Cairo et al 2009) six months after the surgical procedures. Root coverage (RC) is scored zero with no root coverage was obtained (RECH at 6 months is equal to RECH obtained at baseline), three for partial (RECH>0) and six for complete root coverage (RECH=0). Other variables (gingival contour, tissue texture, mucogingival junction alignment and gingival color) are compared to the contra-lateral side and scored up to one point each (zero points if significantly different from contra-lateral side). Thus, this evaluation scale is composed of five independent parameters that result in a total score of 10.

One important patient-related evaluation is the post-surgical pain experienced. In order to quantify the frequence and severity of pain, a visual analog scale (VAS) of pain was employed seven days after the surgical procedure, in which zero meant complete absence of pain and ten the maximum tolerable pain by the patient. Prevalence of pain was documented dichotomously as no pain for VAS scores equal to zero and pain for VAS scores bigger that zero. Severity of pain was quantified by the direct value obtained by the VAS score.

Surgical Procedures were performed by one operator (SK) not involved in clinical data measurements, and patient allocation. Before surgery, each patient was given a single dose of 8mg dexamethasone (EMS, São Paulo, Brasil) to reduce post-surgical edema. Intraoral antisepsis was performed with a 0.12% chlorhexidine rinse (Lacer, Barcelona, Spain). Anesthesia was obtained by regional blocks with 2.0% Mepivacaine with 1:1 00.000 epinephrine (DFL, Rio de Janeiro, Brasil).

Semilunar coronally positioned flap - Conventional approach

The MACRO SLCRF procedure was performed as originally described by Tarnow et al (1986). Briefly, a semilunar incision (SLI) was carried out following the outline of the gingival margin with a 15c surgical blade. This incision ended into the papilla on each interproximal area of the tooth to be treated, but not all the way to the tip of the papilla. At least 2mm of gingiva was preserved on each side of the flap in order to preserve the blood supply. The SLI was curved apically to an extent to guarantee that the apical part of the flap rests on bone after the coronal advancement to cover the root. In order to do that transgingival probing was performed before the incision to determine the position of the bone crest. An intrasulcular incision (ISI) was performed mid-facially. Then, a split-thickness (ST) dissection was performed from the initial incision coronally until connecting to the ISI. The mid-facial tissue was completely released, positioned coronally to the CEJ and held in place against the tooth with a moist gauze pad placed with light pressure, perpendicular to the flap, for five minutes. No sutures were placed, however, a cyanoacrilate adhesive (CAA) was applied over the post-surgical gingival margin and tooth enamel to stabilize the flap.

Semilunar coronally positioned flap - Microsurgical approach

The MICRO SLCRF procedure was performed as described by Bittencourt et al (2006, 2009). Briefly, employing a surgical microscope (DF Vanconcelos, model MC M1232), a SLI was carried out following the outline of the gingival margin with a # 6961 microsurgical blade (Surgistar, California, EUA) under (8x) magnification, the ST dissection, flap advancement and stabilization were performed as descrided above.

Statistical Analysis

All descriptive statistics were expressed as mean +/- standard deviation (SD). Baseline measurements were subjected to inter-group comparisons, and were analyzed by the non-parametric Wilcoxon test or the Chi-square test. Inter-group and intra-group comparisons between baseline and six-month measurements were analyzed by the Wilcoxon test or the Chi-square test. Wilcoxon's signed ranks test was used for intra-group comparisons and the Wilcoxon's rank sums test was used for inter-group comparisons. Statistical significance was set at the 95% probability level (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Presence of bilateral Miller class I gingival recessions (≤ 3mm) exhibiting at least 2mm of keratinized tissue width (WKT) in endodontically-vital maxillary canines or premolars.
* These teeth presented shallow (<3mm) probing depth (PD) without bleeding on probing. Moreover, the elegible individuals demonstrated absence of contraindications for periodontal surgery, and were not being taking medications known to interfere with periodontal tissue health or healing in the preceding 6 months.
* Experimental teeth were free of caries or restorations in the areas to be treated.

Exclusion Criteria:

* Patients with untreated periodontal disease, smokers, subjects with immunosuppressive systemic diseases (i.e., cancer, AIDS, diabetes) were not included in the study.
* Miller class II, III or class IV recession defects, presence of apical radiolucency or caries or restorations in the areas to be treated, and previous lack of cooperation with the maintenance program (as evaluated by unjustified absence from scheduled maintenance visits, continued traumatic tooth brushing technique or faulty plaque control measures).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Root coverage | 6 months
  Distance between the cementum-enamel junction and the gingival margin. Measurements will be performed at baseline (RECH1) and after 6 months (RECH2). The amount of root coverage will be calculated as REC2x100/REC1

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldo B Santana, DDS,MScD,DSc, Principal Investigator — Federal Fluminense University